CLINICAL TRIAL: NCT02783066
Title: Novel Offloading for Diabetic Foot Ulcers With PulseFlow: A Prospective Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Diabetic Boot Company (Industry)
Responsible Party: Principal Investigator, Bijan Najafi, PhD, Professor of Surgery, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: H-37713
Record Dates: First submitted 2016-05-19; First posted 2016-05-26 (Estimated); Results first posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-07

CONDITIONS: Diabetic Foot Ulcer; Offloading
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- "PulseFlow" group (Experimental): Eligible subjects will try a new offloading boot for 4 weeks
  Interventions: Device: Offloading boot: PulseFlow

INTERVENTIONS:
Device: Offloading boot: PulseFlow — A new offloading boot, which may enhance balance, gait, and lower extremity blood flow

SUMMARY:
Diabetic foot ulceration (DFU) is a common and largely preventable complication of diabetes. While most of these ulcers can be treated successfully, some will persist and become infected. Ultimately, nearly one fifth of patients with infected lower-extremity diabetic ulcers will require amputation of the affected limb, resulting in staggering costs for both the patient and the healthcare system. Prevention by identifying people at higher risk is key for better clinical management of such patients. It is not uncommon for patients suffering from diabetes to have concomitant lower extremity edema or venous insufficiency and they subsequently may benefit from graduated compression. However, because of the common association of peripheral arterial disease (PAD) in patients with diabetes, most clinicians are reluctant to apply compressive dressings in fear of exacerbating the symptoms of PAD and possibility of gangrene.

A novel low voltage, battery powered medical device, PulseFlow DF® (The Diabetic Boot Company, Ltd. UK) has endeavored to assist in the treatment of Diabetic Foot Ulcers. The device provides hybrid functionality i.e. mobile air bladder pump at plantar arch and offloading boot. The air bladder inflates to 160 mmHg for approx. 1 second then deflates back to atmospheric pressure, allowing the plantar vessels sufficient time to refill. The offloading boot design holds the foot and lower leg in a position that reduces shear and friction forces and provides a reduction in plantar pressure.

The PulseFlow DF is designed to record how many hours of blood pumping it has delivered. This data will be downloaded at each clinic visit. The boot cannot pump blood around the participant's foot unless fitted correctly and the battery is charged up overnight.

The purpose of this study is to conduct an interventional study study with N=15 diabetic subjects with active foot ulcers to assess whether PulseFlow foot compression device can help improve lower extremity perfusion, whilst improving balance and spatio-temporal parameters of gait.

The key goals of the proposed project are to test whether a specially designed compression device can improve lower extremity perfusion, whilst also simultaneously improving the balance and walking performance. Investigators envision the use of this specially designed offloading device with compression capability will help reduce the incidence of diabetic foot ulcers in high-risk diabetic patients. In addition, investigators assumed the proposed device might enhance daily physical activity as well as walking performance. Investigators will conduct a prospective clinical study to validate these hypotheses. Potential changes in walking and spontaneous daily physical activities will be assessed using validated technologies that include walking analyzer system, balance assessment using body worn sensors, and computerized pressure insoles.

ELIGIBILITY:
Inclusion Criteria:

* 18- 80 years old
* type II diabetes with active plantar ulcer,

Exclusion Criteria:

* Non-ambulatory or unable to stand without help or walk a distance of at least 6 feet without assistance
* Plantar ulcer on arch of the foot
* Patients with PAD (Ankle Brachial Index < 0.5)
* Acute foot fracture
* Heart failure
* Pregnant women
* Patients on immunosuppressive drugs
* Participation in an interventional study in the last 30 days
* Major amputation
* Patients unable or unwilling to participate in all procedures and follow-up evaluations.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-01; Primary Completion 2019-06-30 (Actual); Study Completion 2019-10-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Only de-identified data and associated results will be published in peer-reviewed papers or scientific abstracts

RESULTS

PARTICIPANT FLOW:
Groups:
- "PulseFlow" Group: Eligible subjects will complete gait and balance test with both new offloading boots and standard offloading boots at baseline, and then use new offloading boots for 4 weeks
  Offloading boot : PulseFlow: A new offloading boot, which may enhance balance, gait, and lower extremity blood flow
Period: Overall Study
Arm/Group | "PulseFlow" Group
Started | 16
Completed | 3 (complete 4-week pulseflow offloading wearing test)
Not Completed | 13
Not completed — Withdrawal by Subject | 13

BASELINE CHARACTERISTICS:
Groups:
- "PulseFlow" Group: Eligible subjects will try a new offloading boot for 4 weeks
  Offloading boot : PulseFlow: A new offloading boot, which may enhance balance, gait, and lower extremity blood flow
Arm/Group | "PulseFlow" Group
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 6
  More than one race | 1
  Unknown or Not Reported | 3
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 31.3 (5.9)

OUTCOME MEASURES:

1. Primary Outcome: Lower Extremity Perfusion Change From Baseline to 4 Weeks
Description: Skin perfusion measured in the ankle using Sensilase device. To measure Skin Perfusion Pressure (SPP), a pressure cuff is first automatically inflated to occlude arterial bed blood flow; this is verified by PAD-IQ by determining when perfusion has stopped. The pressure is then automatically released at a controlled rate while the cuff pressure and skin perfusion are measured. A graph displays pressure and perfusion during cuff deflation and indicates the pressure at which skin perfusion is found to return.
Time Frame: baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: percentage of baseline perfusion
Arm/Group | "PulseFlow" Group
Number analyzed (Participants) | 3
percentage of baseline perfusion
  ulcerated | 167 (71)
  contralateral | 75 (51)

2. Primary Outcome: Gait Speed Difference Between Pulseflow Offflaoding and Standard Offloading
Description: the quality of walking while wearing Pulseflow offflaoding compared to standard offloading
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: m/s
Groups:
- "PulseFlow" Group: Eligible subjects will complete gait and balance test with both new offloading boots and standard offloading boots at baseline, and then use new offloading boots for 4 weeks
  PulseFlow: A new offloading boot, which may enhance balance, gait, and lower extremity blood flow
Arm/Group | "PulseFlow" Group
Number analyzed (Participants) | 3
m/s
  Walking speed with Pulse flow offloading | 0.59 (0.20)
  Walking speed with standard offloading | 0.57 (0.20)

3. Secondary Outcome: Adherence
Description: adherence to wear offloading boot by downloading from the study device to a specific developed software. The measure is the mean number of minutes the offloading boot was worn for over the course of 4 weeks
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | "PulseFlow" Group
Number analyzed (Participants) | 3
minutes | 6791 (4914)

4. Secondary Outcome: Wound Size Change From Baseline to 4 Weeks.
Description: measuring the size of the wound (W, L,H)
Time Frame: baselineand and 4 weeks
Measure: Mean (Standard Deviation); unit: percentage of baseline wound area
Arm/Group | "PulseFlow" Group
Number analyzed (Participants) | 3
percentage of baseline wound area | -60 (37)

5. Secondary Outcome: Stride Length Difference Between Pulseflow Offflaoding and Standard Offloading
Description: the quality of walking while wearing Pulseflow offflaoding compared to standard offloading
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: m
Arm/Group | "PulseFlow" Group
Number analyzed (Participants) | 3
m
  standard offlaoding | 0.85 (0.20)
  Pulseflow offlaoding | 0.88 (0.30)

6. Secondary Outcome: Limp Difference Between Pulseflow Offflaoding and Standard Offloading
Description: Limp: the difference in stance percent between right and left feet
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | "PulseFlow" Group
Number analyzed (Participants) | 3
percentage
  standard offlaoding | 4.38 (2.96)
  Pulseflow offlaoding | 2.99 (2.56)

7. Secondary Outcome: Peak Swing Angular Velocity
Description: Angular Velocity of leg swing during walking for each side
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: degree per second
Arm/Group | "PulseFlow" Group
Number analyzed (Participants) | 3
degree per second
  offloaded side of standard offloading | 172.53 (56.85)
  contralateral side of standard offloading | 178.49 (60.31)
  offloaded side of pulseflow offloading | 191.72 (50.52)
  contralateral side of pulseflow offloading | 166.77 (81.65)

8. Secondary Outcome: Ratio of Propulsion Time to Stance Time
Description: Propulsion time and stance time for each stride is caulcated by wearable sensors. The measure is ratio of propulsion time to stance time as percentage value.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: percentage of stance time
Arm/Group | "PulseFlow" Group
Number analyzed (Participants) | 3
percentage of stance time
  offloaded side of standard offloading | 55 (4)
  contralateral side of standard offloading | 60 (8)
  offloaded side of pulseflow offloading | 67 (4)
  contralateral side of pulseflow offloading | 62 (7)

9. Secondary Outcome: Center of Mass Sway While Wearing Standard Offloading Boot
Description: Center of Mass (COM) sway measured by wearable inertial sensors
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | "PulseFlow" Group
Number analyzed (Participants) | 3
cm^2
  double stance with eyes open | 0.18 (0.04)
  double stance with eyes closed | 0.36 (0.04)
  tandem stance with eyes open | 0.38 (0.28)
  tandem stance with eyes closed | 0.74 (0.16)

10. Secondary Outcome: Center of Mass Sway While Wearing Pulseflow Offloading
Description: center of mass sway measured by a wearable inertial sensor
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | "PulseFlow" Group
Number analyzed (Participants) | 3
cm^2
  double stance with eyes open | 0.14 (0.06)
  double stance with eyes closed | 0.46 (0.34)
  tandem stance with eyes open | 0.29 (0.13)
  tandem stance with eyes closed | 0.46 (0.20)

11. Secondary Outcome: Peak Forefoot Pressure
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: Pa
Arm/Group | "PulseFlow" Group
Number analyzed (Participants) | 3
Pa
  offloaded side of standard offloading | 168.7 (156.9)
  contralateral side of standard offloading | 276.7 (105.7)
  offloaded side of pulseflow offloading | 147.0 (114.3)
  contralateral side of pulseflow offloading | 196.9 (84.4)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | "PulseFlow" Group
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-05): https://cdn.clinicaltrials.gov/large-docs/66/NCT02783066/Prot_SAP_000.pdf